CLINICAL TRIAL: NCT00583791
Title: Closure of Muscular Ventricular Septal Defects With The AMPLATZER™ Muscular VSD Occluder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGA-005; G990289
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2016-02

CONDITIONS: Heart Septal Defects, Ventricular
Keywords: muscular; ventricular; septal; defects; VSD
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Main Cohort (Experimental): Device closure with the AMPLATZER Muscular VSD Occluder for patients with muscular ventricular septal defects which are hemodynamically significant and are either isolated or present in conjunction with other congenital heart defects.
  Interventions: Device: Device closure with the AMPLATZER Muscular VSD Occluder

INTERVENTIONS:
Device: Device closure with the AMPLATZER Muscular VSD Occluder — Device: AMPLATZER Muscular VSD Occluder

SUMMARY:
The objective is to investigate the safety of the AMPLATZER Muscular VSD Occluder for the treatment of muscular ventricular septal defects, which are hemodynamically significant and are either isolated or in conjunction with other congenital heart defects in infants and children.

DETAILED DESCRIPTION:
The objective of this feasibility study is to investigate the safety of the AMPLATZER Muscular VSD Occluder for the treatment of muscular ventricular septal defects, which are hemodynamically significant and are either isolated or in conjunction with other congenital heart defects in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemodynamically significant muscular VSD's (demonstrated by echocardiography or angiography), either isolated or in conjunction with other congenital heart defects
* Age < 18 years old

Exclusion Criteria:

* Less than 4 mm distance from the semilunar (aortic and pulmonary) and atrioventricular valves (mitral and tricuspid)
* Patients with severely increased pulmonary vascular resistance above 7 woods units and a right-to-left shunt and documented irreversible pulmonary vascular disease
* Patients with perimembranous (close to the aortic valve) VSD
* Patients < 3 kg
* Patients with sepsis (local/generalized)
* Patients with gastritis, gastric ulcer, duodenal ulcer, bleeding disorders etc. and other contraindications to aspirin therapy unless other anti-platelet agents can be administered for 6 months
* Inability to obtain informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2000-07; Primary Completion 2008-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Levi, MD, Principal Investigator — University of California, Los Angeles
Locations (11):
- United States (11):
  - Children's Hospital, Denver, Colorado
  - Arnold Palmer Hospital, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbus Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Cohort: Treatment of muscular VSDs (ventricular septal defects) which are hemodynamically significant and are either isolated or present in conjunction with other congenital heart defects.
Period: Overall Study
Arm/Group | Main Cohort
Started | 91
Completed | 18
Not Completed | 73
Not completed — Other | 67
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Groups:
- Main Cohort: Patients with muscular VSDs that are hemodynamically significant and are either isolated or present in conjunction with other congenital heart defects.
Arm/Group | Main Cohort
Number analyzed (Participants) | 91
Age, Continuous [Mean (Full Range); unit: years] | 6.66 [0.03 to 54.05]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 91

OUTCOME MEASURES:

1. Primary Outcome: Closure of Muscular Ventricular Septal Defects
Description: Closure of muscular ventricular septal defect with the AMPLATZER Muscular VSD Occluder
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Main Cohort
Number analyzed (Participants) | 91
participants | 91

ADVERSE EVENTS:
Arm/Group | Main Cohort
All-Cause Mortality (participants affected / at risk) | 6/91
Serious Adverse Events (participants affected / at risk) | 29/91
Other Adverse Events (participants affected / at risk) | 74/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=91)
AE Code Not Specified (General disorders) | 1 (1)
Anemias (General disorders) | 1 (1)
Anemias Caused By Blood Loss (General disorders) | 2 (2)
Arterial Pulse Loss (General disorders) | 2 (2)
Blood Loss (General disorders) | 5 (5)
Blood Transfusion (General disorders) | 5 (5)
Bradycardia (General disorders) | 1 (1)
Cardiac Arrest (General disorders) | 2 (2)
Cardiac Perforation (General disorders) | 2 (2)
Cardiac Surgery (General disorders) | 1 (1)
Cardiomyopathy (General disorders) | 1 (1)
Death1 (General disorders) | 3 (3)
Delivery System Failure (General disorders) | 2 (2)
Device Collapse2 (General disorders) | 1 (1)
Device Embolization3 (General disorders) | 2 (2)
Dual Pacemaker (General disorders) | 1 (1)
Encephalopathy (General disorders) | 1 (1)
Hematoma (General disorders) | 1 (1)
Hemostasis and Coagulation Disorders (General disorders) | 1 (1)
Hypotension (General disorders) | 5 (5)
Mobitz II Block (General disorders) | 1 (1)
Paroxysmal Ventricular Tachycardia (General disorders) | 1 (1)
Poor Device Position (General disorders) | 1 (1)
Seizures (General disorders) | 1 (1)
Stroke (General disorders) | 2 (2)
Subaortic Stenosis (General disorders) | 2 (4)
Third Degree Heart Block (Complete Heart Block) (General disorders) | 3 (3)
Vocal cord paralysis (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=91)
AE Code Not Specified (General disorders) | 1 (1)
Acidosis (General disorders) | 1 (1)
Acute Bronchitis (General disorders) | 1 (1)
Acute Erosive Gastritis (General disorders) | 1 (1)
Acute Otitis Media (General disorders) | 2 (3)
Acute Pancreatitis (General disorders) | 2 (2)
Acute Pharyngitis (General disorders) | 1 (1)
Anemias (General disorders) | 2 (2)
Anemias Caused By Blood Loss (General disorders) | 2 (2)
Anemias Caused By Deficient Erythropoiesis (General disorders) | 1 (1)
Anesthesia Reaction (General disorders) | 1 (1)
Arrhythmias (General disorders) | 2 (2)
Arterial Pulse Loss (General disorders) | 2 (2)
Asthma (General disorders) | 4 (4)
Atelectasis (General disorders) | 8 (8)
Atopic Dermatitis (General disorders) | 1 (1)
Atrial Fibrillation (General disorders) | 1 (1)
Atrial Flutter (General disorders) | 1 (1)
Bacteremia (General disorders) | 4 (4)
Bacterial Infections (General disorders) | 4 (6)
Biventricular Hypertrophy/Combined Ventricular Hypertrophy (General disorders) | 1 (1)
Blood Loss (General disorders) | 5 (5)
Blood Transfusion (General disorders) | 6 (6)
Bradycardia (General disorders) | 4 (4)
Broad QRS Complex Arrhythmias (General disorders) | 1 (1)
Bronchomalacia (General disorders) | 1 (1)
Bruise/Purpura Simplex (General disorders) | 1 (1)
CVVH (Continuous Veno Venous Hemofiltration) (General disorders) | 1 (1)
Cardiac Arrest (General disorders) | 2 (2)
Cardiac Perforation (General disorders) | 2 (2)
Cardiac Cath (General disorders) | 1 (1)
Cardiac Surgery (General disorders) | 13 (14)
Cardiomyopathy (General disorders) | 3 (3)
Cellulitis (General disorders) | 1 (1)
Chest Pain (General disorders) | 4 (5)
Cholecystitis (General disorders) | 1 (1)
Chronic Recurrent Drainage/Oozing (General disorders) | 1 (1)
Circumcision (General disorders) | 1 (1)
Coarctation of Aorta (General disorders) | 1 (1)
Cobra Formation (General disorders) | 1 (1)
Common Cold/Upper Respiratory Tract Infection (General disorders) | 9 (16)
Congestive Heart Failure (General disorders) | 2 (2)
Conjunctivitis (General disorders) | 1 (1)
Cough (General disorders) | 2 (2)
Croup (General disorders) | 2 (2)
Cyanosis (General disorders) | 1 (1)
Death* (General disorders) | 4 (4)
Dehydration (General disorders) | 2 (2)
Delivery System Failure (General disorders) | 4 (4)
Device Collapse (General disorders) | 1 (1)
Device Embolization (General disorders) | 2 (2)
Diabetes Mellitus (General disorders) | 1 (1)
Dizziness (General disorders) | 3 (3)
Dual Pacemaker (General disorders) | 2 (3)
Dyspnea (General disorders) | 4 (4)
Edema (General disorders) | 3 (3)
Elective Surgery (General disorders) | 2 (3)
Elective Adenoidectomy with Tympanostomy Tubes (General disorders) | 1 (1)
Encephalopathy (General disorders) | 1 (1)
Fever (General disorders) | 4 (7)
First Degree Heart/AV Block/Cardiac Arrhythmia - 1st Degree AV Block (General disorders) | 1 (1)
Foreign Bodies (General disorders) | 2 (2)
Fracture (General disorders) | 1 (1)
Functional Vomiting (General disorders) | 1 (1)
Fungal Pneumonia (General disorders) | 1 (1)
Gastroesophageal Reflux Disease (General disorders) | 4 (4)
Gastrointestinal Bleeding (General disorders) | 1 (1)
Gastrostomy Tube (General disorders) | 1 (1)
Headache (General disorders) | 3 (3)
Hematoma (General disorders) | 4 (4)
Hematoma of the Groin (General disorders) | 2 (2)
Hematuria (General disorders) | 1 (1)
Hemostasis and Coagulation Disorders (General disorders) | 2 (2)
Hyperglycemia (General disorders) | 1 (1)
Hypotension (General disorders) | 10 (10)
Incomplete Right Bundle Branch Block (General disorders) | 2 (2)
Ingestion (General disorders) | 1 (1)
Interventricular Conduction Delay (General disorders) | 1 (1)
Junctional Escape Beat (General disorders) | 1 (1)
Junctional Escape Rhythm/Intermittent Junctional Rhythm (General disorders) | 2 (2)
Lacerations (General disorders) | 1 (2)
Left Ventricular Hypertrophy (General disorders) | 1 (1)
Liver Enlargement (General disorders) | 1 (1)
Meatal Stenosis (General disorders) | 1 (1)
Memory Loss (General disorders) | 1 (1)
Metabolic Alkalosis (General disorders) | 1 (1)
Migraine (General disorders) | 1 (1)
Mild Mitral Valve Regurgitation (General disorders) | 1 (1)
Mild Tricuspid Regurgitation (General disorders) | 3 (3)
Miscellaneous Infections (General disorders) | 2 (2)
Mitral Valve Regurgitation/Mitral Insufficiency (General disorders) | 1 (1)
Mobitz II Block (General disorders) | 5 (5)
Moderate Tricuspid Regurgitation (General disorders) | 1 (1)
Musculoskeletal Pain (General disorders) | 1 (1)
Myalgias (General disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Nonspecific Intraventricular Conduction Defects (General disorders) | 3 (3)
Nose Bleed (General disorders) | 1 (1)
Other (General disorders) | 1 (1)
Otitis Media (General disorders) | 1 (1)
Pallor (General disorders) | 1 (1)
Palpitations (General disorders) | 2 (2)
Paroxysmal Junctional Tachycardia (General disorders) | 1 (1)
Paroxysmal Ventricular Tachycardia (General disorders) | 3 (3)
Pericardial Effusion (General disorders) | 4 (5)
Pharyngitis (General disorders) | 2 (2)
Pleural Effusions (General disorders) | 3 (3)
Pleuropericardial Fluid (General disorders) | 1 (1)
Pneumonia (General disorders) | 4 (6)
Pneumonia Caused By Gram-Negative Bacilli (General disorders) | 1 (1)
Pneumothorax (General disorders) | 1 (1)
Poor Device Position (General disorders) | 1 (1)
Premature Atrial Beat (General disorders) | 1 (1)
Premature Ventricular Contraction (General disorders) | 2 (2)
Pulmonary Congestion (General disorders) | 1 (1)
Pulmonary Hemorrhage (General disorders) | 1 (1)
Pulmonary Hypertension (General disorders) | 1 (1)
Pulmonary Stenosis (General disorders) | 1 (1)
Pulmonary Edema (General disorders) | 6 (7)
Rash (General disorders) | 3 (3)
Renal Failure (General disorders) | 1 (1)
Respiratory Synctial Virus Infection (RSV) (General disorders) | 3 (3)
Right Bundle Branch Block/Complete Right Bundle Branch Block (General disorders) | 11 (13)
Right Ventricular Hypertrophy (General disorders) | 1 (1)
Scoliosis (General disorders) | 1 (1)
Seizure/Convulsions/Epilepsy (General disorders) | 1 (1)
Seizures (General disorders) | 3 (3)
Sinusitis (General disorders) | 5 (6)
Stridor (General disorders) | 1 (1)
Stroke (General disorders) | 2 (2)
Subaortic Stenosis (General disorders) | 2 (4)
Subglottic Edema 2 to Prolonged Intubation (General disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Tachypnea (General disorders) | 1 (1)
Third Degree Heart Block (Complete Heart Block) (General disorders) | 5 (6)
Trace Tricuspid Regurgitation (Tricuspid Incompetence or Ins) (General disorders) | 1 (1)
Tracheostomy (General disorders) | 2 (2)
Trigeminy (General disorders) | 1 (1)
Urinary Tract Infections (General disorders) | 1 (1)
Vascular Congestion (General disorders) | 1 (1)
Venous Thrombosis (General disorders) | 1 (1)
Ventricular Escape Rhythm (General disorders) | 1 (1)
Viral Gastroenteritis (General disorders) | 3 (4)
Viral Pneumonia (General disorders) | 1 (1)
Vocal Cord Paralysis (General disorders) | 1 (1)
Vomiting (General disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No